CLINICAL TRIAL: NCT05258526
Title: Home Based Exercise for Patients With Breast or Prostate Cancer During Treatment: a Feasibility Trial (The BENEFIT-CA Study)
Brief Title: Home Based Exercise for Patients With Breast or Prostate Cancer (The BENEFIT-CA Study)
Acronym: BENEFIT-CA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0262
Record Dates: First submitted 2022-02-07; First posted 2022-02-28 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer; Prostate Cancer
Keywords: Cancer; Feasibility trial; Physical activity; Home based exercise; Trial adherence
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: This a feasibility trial to assess a home-based exercise intervention individuals with breast or prostate cancer during treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home-based exercise program (Experimental): This is a single study arm consisting of a home-based exercise program for individuals with breast or prostate cancer during active treatment.
  Interventions: Other: Home based exercise training

INTERVENTIONS:
Other: Home based exercise training — The intervention will be based on a remote approach, lasting 12 weeks. The training routine will consist of aerobic (walking), muscle strengthening and stretching exercises, with a frequency of three days per week. The contents related to the exercise prescription will be made available by phone call, text messages and short videos for exercise demonstration.

SUMMARY:
The purpose of this trial is to evaluate the feasibility of a home based exercise program for individuals with breast or prostate cancer patients undergoing active treatment.

DETAILED DESCRIPTION:
This feasibility trial aims to assess a home-based exercise program, including a 3-month intervention of structured physical activity and health education for individuals with breast or prostate cancer. The main objective of this trial is to assess the adherence of cancer patients to a program of structured exercise, mixed with a health education approach, implemented and accompanied in a remote approach.

The data collection will include variables related to: (a) recruitment and retentions rates; (b) attendance to exercise sessions; (c) fatigue and quality of life levels; (d) functional capacity levels; (e) adverse events related or not to the study; (f) patient selected outcomes.

ELIGIBILITY:
Inclusion Criteria:

* eighteen years old minimum;
* be living in Porto Alegre or metropolitan region;
* breast cancer stage 0 - III OR
* localized prostate cancer;
* undergoing hormonal treatment / manipulation in isolation or combined with other therapies three months prior to the entrance in the study;
* hormonal therapy / manipulation planned to be active throughout the study duration;
* not engaged in any exercise training for more than once a week for the past 6 months;
* in case of previous surgical procedure, the patient must have medical clearance at the moment of the contact to begin the study or be cleared to do so in the near future (up to two weeks).

Exclusion Criteria:

* metastatic phase / progression of the disease or active regional location prior to beginning of the study;
* inability to understand the terms and conditions of study due to language, hearing, cognitive or severe psychiatric issues;
* another family member, who lives at the same residence, participating in the study;
* planning to move or major absence (more than two weeks) during the study;
* history of cardiovascular disease (except controlled hypertension) or severe cardiopulmonary disease, as well as history of heart attack, revascularization procedures, profound venous thrombosis, encephalic vascular accident (brain stroke) or pulmonary embolism in the past twelve months;
* chronic pulmonary disease that requires oxygen or corticosteroid therapy;
* kidney disease with or that is going to begin the use of dialysis or waiting for a kidney transplant;
* severe nausea, anorexia or any other condition which does not allow to perform physical exercise;
* medical contraindication to exercise training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The trial is designed for female breast cancer patients and male prostate cancer patients.
Enrollment: 80 (Estimated)
Dates: Start 2022-04-07 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Trial adherence | Up to12 weeks.
  Proportion of self-reported exercise episodes (out of 36 episodes, total) during the study.

SECONDARY OUTCOMES:
Recruitment yields | Up to 8 weeks before allocation to the study intervention.
  Proportion of included participants (who signed the informed consent) in relation to the total number of screened individuals for eligibility.
Adverse events throughout the study | Up to 12 weeks.
  Self-reported adverse events, related or not to the study. These measures will be mostly received by phone calls or text messaging.

OTHER OUTCOMES:
Fatigue levels at baseline and at the end of the study | Baseline; Week 12.
  Fatigue scores using specific questionnaires of Functional Assessment of Cancer Therapy (FACT questionnaire) for breast or prostate cancer patients.
Quality of life, based on the Functional Assessment of Cancer Therapy (FACT questionnaire) | Baseline; Week 12.
  Quality of life scores using specific questionnaires of FACT (Functional Assessment of Cancer Therapy) for breast or prostate cancer patients.
Walking capacity | Baseline; Week 12.
  Total distance (in meters) performed during the six minute walk test.
Handgrip strength | Baseline; Week 12.
  Maximum strength (in kgf) achieved by both hands in a handgrip test using a hand dynamometer.
Abdominal circumference | Baseline; Week 12.
  Anthropometric measure of the highest abdominal circumference, using a metallic measuring tape.
Physical activity levels | Single assessment at baseline.
  Physical activity calculated in minutes and intensity per week, of physical activity using the International Physical Activity Questionnaire (IPAQ).
Patient selected outcomes | Week 12.
  Through the development of the study, participants will be asked to engage in a focal group to discuss outcomes relevant to be assessed in trials with exercise interventions targeted for patients with breast or prostate cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Umpierre de Moraes, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Files will be as de-identified as possible before public data sharing. After data protection and data handling routines, de-identified data will be readily available to all project contributors. We consider research data gathered from data collection from research participants pertains primarily to these individuals. Therefore, all individual data will be available to their owners throughout the project. Structured data that will result from this research project will pertain to the PI (Daniel Umpierre), who will be responsible for data integrity, and to the institution (Hospital de Clinicas de Porto Alegre).
  The specific structure for data sharing as well as plataforms are still to be defined. As soon, we define the remaining details of our data sharing strategy the IPD plan will be updated.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Due to space and management constraints, we are planning:
  1. To retain and store project documentation (informed consents, IRB communication, subjects' communication) for at least 10 years after the study completion (anticipated time: up to 2033).
  2. To retain and share project resources (instruments, intervention materials) as long as public repositories (e.g., Zenodo, OSF, figshare) provide sharing services at no cost.
  3. To retain and share datasets as long as public repositories (e.g., Zenodo, OSF, figshare) provide sharing services at no cost.
Access Criteria: All the files will be password-protected and only investigators or data managers designated to use the files will be given access. Different passwords will be used for different users, which allows auditing to be made more easily. Although we do not plan to request justification to release the datasets, we do plan to share the data in a controlled approach. Therefore, once the datasets are made available at the Zenodo.org platform, only registered users will be able to download files. This procedure allows us to keep a record of data requests.
URL: https://osf.io/gw2x6/

REFERENCES:
- [Derived] da Silva LXN, Leite JS, Ignacio AC, Massierer FD, Pfeifer LO, Dos Santos Cardoso LA, Alano TS, Umpierre D. The "home-based exercise for breast and prostate cancer patients during treatment-a feasibility trial" (BENEFIT CA trial): rationale and methodological protocol. Pilot Feasibility Stud. 2023 Sep 26;9(1):165. doi: 10.1186/s40814-023-01393-0. PMID 37752564